CLINICAL TRIAL: NCT06014671
Title: The Effect of Interpersonal Psychotherapy on Quality of Life Among People Living With HIVAIDS at Mettu Karl Referral and Bedele Hospital, Southwest Ethiopia, 2022: A Quasi-experimental Study
Brief Title: The Effect of Interpersonal Psychotherapy on Quality of Life Among People Living With HIVAIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mattu University (Other)
Responsible Party: Principal Investigator, Zakir Abdu, Assistant Professor of Psychiatry, Mattu University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHS/54/2014
Record Dates: First submitted 2023-08-14; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Breif Description: Patients' Quality of Life of
MeSH Terms: interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): intervention group were took interpersonal psychotherapy
  Interventions: Behavioral: Interpersonal Psychotherapy
- Control group (Experimental): control group didn't took interpersonal psychotherapy
  Interventions: Behavioral: Interpersonal Psychotherapy

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy — Intervention Group were took interpersonal psychotherapy

SUMMARY:
Quality of life (QOL) is a significant importance for people living with HIV/AIDS by modifying the adverse psychosocial consequences that accompany the disease. In Ethiopia, interpersonal psychotherapy (IPT) has never been tried for people living with HIV/AIDS for quality of life. The objective of the study was to assess the effects of interpersonal psychotherapy on quality of life among PLWHA at Mettu Karl referral and Bedele hospital, southwest Ethiopia, 2022.

ELIGIBILITY:
Inclusion Criteria:

* PLWHA who were 18 years of age or above were included in the study

Exclusion Criteria:

* PLWHA who are either currently or previously used IPT and acute physical or mental disturbances will be excluded

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
The effect of Interpersonal Psychotherapy on quality of life among people living with HIVAIDS | two months
  Quality of Life measured by World Health Organization Health Related Quality of Life (WHOQOL- BREF).

CONTACTS AND LOCATIONS:
Locations (1):
- Mattu University, Addis Ababa, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
researchers need information could get it
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: at any time
Access Criteria: with formal letter and justification